CLINICAL TRIAL: NCT04769037
Title: "SINT1A" - Supplementation With B. Infantis for Mitigation of Type 1 Diabetes Autoimmunity - A Study of the Global Platform for the Prevention of Autoimmune Diabetes ("GPPAD")
Brief Title: Supplementation With B. Infantis for Mitigation of Type 1 Diabetes Autoimmunity
Acronym: SINT1A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helmholtz Zentrum München (Industry)
Collaborators: Technical University of Munich (Other); Kinderkrankenhaus auf der Bult (Other); University Hospital Carl Gustav Carus (Other); Skane University Hospital (Other); Universitaire Ziekenhuizen KU Leuven (Other); Medical University of Warsaw (Other); Cambridge Biomedical Campus, Cambridge, UK (Unknown); Royal Victoria Infirmary, Newcastle upon Tyne, UK (Unknown)
Responsible Party: Principal Investigator, Anette-Gabriele Ziegler, Director - Institute of Diabetes Research, Helmholtz Zentrum München
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPPAD-04
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes autoimmunity; celiac autoimmunity; respiratory infections; allergy; prevention; probiotic; B. infantis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Respiratory Tract Infections; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B. infantis (Active Comparator): Activated B. infantis EVC001; Bifidobacterium longum subsp. infantis; 8 x 109 colony forming units (CFU) per day
  Interventions: Dietary Supplement: B. infantis
- Placebo (Placebo Comparator): Lactose identical in appearance and taste to the active supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. infantis — Activated B. infantis EVC001; Bifidobacterium longum subsp. infantis; 8 x 109 colony forming units (CFU) per day
  Arms: B. infantis
Dietary Supplement: Placebo — Lactose identical in appearance and taste to the active supplement
  Arms: Placebo

SUMMARY:
Investigator initiated, randomised, placebo-controlled, double-blind, multi-centre primary intervention study to assess whether daily administration of B. infantis EVC001 from age 7 days to 6 weeks (+14 days) until age 12 months (+ 14 days) to children with elevated genetic risk for type 1 diabetes reduces the cumulative incidence of beta-cell autoantibodies in childhood.

DETAILED DESCRIPTION:
The GPPAD-04 SINT1A study will evaluate whether early, regular supplementation with a daily dose of a probiotic can reduce the risk of developing beta-cell autoimmunity in children identified by GPPAD-02 as being genetically predisposed to developing type 1 diabetes. Children will be enrolled at age 7 days to 6 weeks (+14 days) and the study product (B. infantis EVC001 or Placebo) will be administered orally once per day from enrollment until age 12 months (+14 days).

The hypotheses is that administration of B. infantis may have a positive influence on the intestinal flora and thus have a regulating effect on the immune system. The study is designed to investigate whether pathogenic immune reactions as in type 1 diabetes but also in other diseases, such as celiac disease, can be reduced and if the disease can be prevented.

Children will be followed until age 3.5 - 6.5 years (2.5 - 5.5 years after end of treatment).

Throughout the study data will be collected by regular study visits, phone calls with the families and electronic questionaires.

Blood samples will be collected to investigate glucose, HbA1c, beta-cell autoantibodies, transglutaminase antibodies, vaccine responses, genetic susceptibility and mechanistic markers. Stool samples will be collected for further assessments such as colonization,microbiome, pH and calprotectin.

Exploratory outcomes (allergy, vaccine responses, stool microbiome, blood metabolomics, stool pH and calprotectin or site specific ancillary measurements) may be assessed or in part assessed on a portion of the participants after unblinding the study. They may not necessarily be included in the primary outcome analysis and publication.

GPPAD is committed to sharing of data in compliance with all applicable European and GPPAD Consortium Member State, Data Protection and Privacy Protection laws, rules and regulations.

Pseudonymized data of the GPPAD-04 SINT1A study will be available to the scientific community after the publication of the trial analysis, which is anticipated in 2028. The SINT1A data will be available upon request.

ELIGIBILITY:
Inclusion Criteria:

1. Infants between the ages of 7 days and 6 weeks (+14 days in case of illness or COVID-19 related issues or unexpected delay in result reporting) at the time of randomisation.
2. A 10% or higher genetic risk to develop multiple beta-cell autoantibodies by age 6 years:

   1. For infants without a first-degree family history of type 1 diabetes, high genetic risk is defined as a DR3/DR4-DQ8 or DR4-DQ8/DR4-DQ8 genotype and a genetic risk score that is in the upper 25th centile (>14.4) or a DR3/DR4-DQ8 genotype with a GRS between the upper 50th (14.0) and 25th centile and a GG genotype at the rs3763305 SNP. These represent around 1% of all newborns.
   2. For infants with a first-degree family history of type 1 diabetes, high genetic risk is defined as having HLA DR4 and DQ8, and none of the following protective alleles: DRB1*1501, DQB1*0503, DRB1*1303. These represent around 30% of infants with a first-degree family history of T1D.
3. Written informed consent signed by the custodial parent(s).-

Exclusion Criteria:

1. Any medical condition, concomitant disease or treatment that may interfere with the assessments or may jeopardize the participant's safe participation in the study, as judged by the Investigators.
2. Preterm delivery < 36 weeks of gestation.
3. Proven immunodeficiency.
4. Any condition that could be associated with poor compliance.5. Diagnosis of diabetes at the time of recruitment

Ages: 7 Days to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1149 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Persistent confirmed multiple beta-cell autoantibodies | Through study completion, up to 6.5 years
  Persistent confirmed multiple beta-cell autoantibodies is defined as confirmed IAA, confirmed GADA, confirmed IA-2A, or confirmed ZnT8A in two consecutive samples, AND a confirmed second antibody from these four antibodies in one sample.
  The primary outcome is the elapsed time from the random treatment assignment to the first confirmed autoantibody positive sample used in defining the persistent confirmed multiple beta-cell autoantibody positive status. Diabetes in the absence of multiple beta-cell autoantibodies is also considered as a primary outcome endpoint, and in this case, the date of diagnosis is the time of the end point.

SECONDARY OUTCOMES:
Persistent confirmed beta-cell autoantibodies | Through study completion, up to 6.5 years
  Any persistent confirmed beta-cell autoantibody, defined as at least one confirmed autoantibody in two consecutive samples, including IAA, GADA, IA-2A or ZnT8A
Diabetes | Through study completion, up to 6.5 years
  Criteria for T1D onset are, as defined by the American Diabetes Association (ADA), based on glucose testing, or the presence of unequivocal hyperglycaemia with acute metabolic decompensation (diabetic ketoacidosis).
Transglutaminase antibodies | Through study completion, up to 6.5 years
  Transglutaminase antibodies defined as persistent in two consecutive samples
Respiratory infection rate | 1 year
  Respiratory infection rate in first year of life during supplementation
Measurement of Safety parameters | from Baseline until 30 days after end of supplementation
  Adverse Events and Serious Adverse Events will be captured until 30 days after the last administration of the food product.
  Local and systemic adverse effects will be elicited by direct questioning of the participant or parent. Systemic effects will be sought by questioning about any untoward symptoms or signs, and graded as mild, moderate, severe, life-threatening or death according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

OTHER OUTCOMES:
Allergy | Through study completion, up to 6.5 years
  Participant's parents will be asked to complete questionnaires to obtain information about allergies every 12 months. Analyses will compare the B. infantis supplementation and placebo groups for the frequency of allergy and allergy sub-groups as defined form the yearly questionnaires.
Antibody response (IgG titres) to vaccines | at age 6 months (rotavirus) and at age 2 years (MMR)
  Information about rotavirus and MMR vaccination will be collected from parents and antibody response (IgG titers) will be measured centrally.
Alterations of the gut microbiome or blood metabolome | from baseline to age 12 months
  Exploratory analyses will examine the associations between B. infantis supplementation and mouth and stool organisms (microbiome), and blood markers such as the metabolome.
Stool pH | at age 6 months
  Stool pH levels will be compared between B. infantis supplementation and placebo groups in a subset of children
Stool calprotectin | at age 6 months
  Stool calprotectin levels will be compared between B. infantis supplementation and placebo groups in a subset of children

CONTACTS AND LOCATIONS:
Locations (8):
- University Hospitals Leuven Faculty of Medicine, Catholic University of Leuven, Leuven, Belgium
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus Technische Universität Dresden, Dresden
  - AUF DER BULT, Kinder- und Jugendkrankenhaus, Hanover
  - Institute of Diabetes Research, Helmholtz Zentrum Munich, Germany, and Forschergruppe Diabetes, Technical University Munich (TUM), School of Medicine, Klinikum rechts der Isar, Munich
- Department of Paediatrics Medical University of Warsaw, Warsaw, Poland
- Lund University, Skane University Hospital SUS, Malmo, Sweden
- United Kingdom (2):
  - University Department of Paediatrics, Cambridge Biomedical Campus, Cambridge
  - Royal Victoria Infirmary, Newcastle upon Tyne, Newcastle

IPD SHARING:
Plan to Share IPD: No
GPPAD is committed to sharing of data in compliance with all applicable European and GPPAD Consortium Member State, Data Protection and Privacy Protection laws, rules and regulations.
  Pseudonymized data of the GPPAD-04 SINT1A study will be available to the scientific community after the publication of the trial analysis, which is anticipated in 2028. The SINT1A data will be available upon request.

REFERENCES:
- [Derived] Ziegler AG, Arnolds S, Kolln A, Achenbach P, Berner R, Bonifacio E, Casteels K, Elding Larsson H, Gundert M, Hasford J, Kordonouri O, Lundgren M, Oltarzewski M, Pekalski ML, Pfirrmann M, Snape MD, Szypowska A, Todd JA; GPPAD STUDY GROUP. Supplementation with Bifidobacterium longum subspecies infantis EVC001 for mitigation of type 1 diabetes autoimmunity: the GPPAD-SINT1A randomised controlled trial protocol. BMJ Open. 2021 Nov 9;11(11):e052449. doi: 10.1136/bmjopen-2021-052449. PMID 34753762
- See also: Related Info — https://www.gppad.org/en/